CLINICAL TRIAL: NCT03799965
Title: Investigation of the Effect of Enhanced Recovery After Surgery (ERAS) Program on Postoperative Results of Patients Operated for Open Heart Surgery
Brief Title: The Effect of Advanced Improvement Program (ERAS) on Postoperative Outcomes in Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Collaborators: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ipek Yakin Duzyol, specialist doctor, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: KUGOKAEK 2017/369
Record Dates: First submitted 2018-12-30; First posted 2019-01-10 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Enhanced Recovery After Surgery; Open Heart Surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS protocol are evaluated (Active Comparator): * It is to compare the durations of stay in the intensive care unit and in hospital
  * It is to compare the incidences of complications of the groups
  Interventions: Other: ERAS (Enhanced Recovery After Surgery ) are evaluated
- ERAS protocol are not evaluated (Active Comparator): * It is to compare the durations of stay in the intensive care unit and in hospital
  * It is to compare the incidences of complications of the groups
  Interventions: Other: ERAS are not evaluated

INTERVENTIONS:
Other: ERAS (Enhanced Recovery After Surgery ) are evaluated — In this arm ERAS( Enhanced Recovery After Surgery) protocol will be inserted.The findings regarding the patients under ERAS protocol are evaluated based on evidence.
  Arms: ERAS protocol are evaluated
Other: ERAS are not evaluated — In this arm ERAS( Enhanced Recovery After Surgery) protocol will not be inserted.The findings regarding the patients under ERAS protocol are evaluated based on evidence.
  Arms: ERAS protocol are not evaluated

SUMMARY:
Investigation of the effect of Enhanced Recovery After Surgery (ERAS) program on postoperative results of patients operated for open heart surgery.

DETAILED DESCRIPTION:
The ERAS protocol, also known as evidence based "fast-track surgery" (FTS), is an evidence based combination of findings regarding suggestions for patient care on various levels of the perioperative period, which work in synergy for accelerating the postoperative recovery period. It has been used sucessfully for many surgical disciplines, primarily colorectal surgery, since it was first reported in 1997. However, there is a significant insufficiency of this patient oriented rehabilitation program regarding cardiovascular surgeries. This study is to compare the postoperative follow up periods of patients with ERAS protocol and patients with standard protocol who were both operated for cardiac surgery.

Following approval of the local ethics committee, 210 patients who are operated for elective cardiac surgery are enrolled in this prospective randomized clinical trial. The patients who are not applied the ERAS protocol are evaluated in the control group (n=51). The findings regarding the patients under ERAS protocol are evaluated based on evidence. Our primary is to compare the durations of stay in the intensive care unit and in hospital; our secondary is to compare the incidences of complications of the groups. The demographic data, operative measurements, complication rates, the amounts of perioperative bleeding and drainage and the duration of stay in the intensive care unit and hospital are recorded.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old;
* Patients undergoing elective open heart surgery (cardiopulmonarybiasis, aortic and mitral valve replacement);
* ASA III ;
* Patients with informed consent for the study.

Exclusion Criteria:

* Patients who refuse to participate in the study;
* Patients under emergency conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
durations of stay | 24 hours
  compare the durations of stay in the intensive care unit and in hospital
complications | 24 hours
  compare the incidences of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Emine yurt, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided